CLINICAL TRIAL: NCT06884345
Title: Safety and Efficacy of METR-NK Cells Combined With Solantinib Neoadjuvant Therapy in HRD+ Advanced Epithelial Ovarian Cancer: a Single-arm, Single-center, Exploratory Clinical Study
Brief Title: METR-NK Cells in Combination With Anti-angiogenic Neoadjuvant Therapy for Advanced Epithelial Ovarian Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Anhui Provincial Cancer Hospital (Other)
Responsible Party: Principal Investigator, Bai-Rong Xia, Director of Gynecological Surgery, Anhui Provincial Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025 NO.01
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental)
  Interventions: Drug: METR-NK cells combined with Solvatinib

INTERVENTIONS:
Drug: METR-NK cells combined with Solvatinib — Sorafenib 250mg po qd, 3 weeks as a course, a total of 3 courses, the drug was stopped 3 weeks before cytoreduction of intermediate tumor.
  Dilute METR - 200 mL of NK cells in 37 ℃ 1500 mL of 0.9% sodium chloride physiological saline, intraperitoneal infusion, flow rate > 150 drops/min, each METR - venous back to the throughput of NK cells is lower than 2 x 107 cells/kg, abdominal cavity to throughput of no less than 4 x 107 cells/kg, Three days of continuous infusion was taken as a course of treatment, and four courses of continuous infusion (the first course of infusion did not use METR-NK cells) were given, with an interval of 14 days for each course. The position was switched every 15 min after the completion of each infusion to ensure uniform distribution of cells to the tumor surface.

SUMMARY:
To further evaluate and observe the efficacy and safety of solantinib combined with METR-NK neoadjuvant therapy for advanced epithelial ovarian cancer in patients with advanced epithelial ovarian cancer by using solantinib combined with METR-NK neoadjuvant therapy

DETAILED DESCRIPTION:
Sorafenib 250mg po qd, 3 weeks as a course, a total of 3 courses. Dilute METR - 200 mL of NK cells in 37 ℃ 1500 mL of 0.9% sodium chloride physiological saline, intraperitoneal infusion, flow rate > 150 drops/min, each METR - venous back to the throughput of NK cells is lower than 2 x 107 cells/kg, abdominal cavity to throughput of no less than 4 x 107 cells/kg, Three consecutive reinfusion days were taken as a course, and four consecutive reinfusion courses were given, with an interval of 14 days between each course. The position was changed every 15 min after the end of each infusion to ensure that the cells were evenly distributed to the tumor surface to achieve the therapeutic effect.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old (≥18, ≤70);
* Open surgery, laparoscopic surgery or coarse needle puncture biopsy and pathology confirmed late in the center of the local laboratory (FIGO IIIC/IV) high grade serous ovarian cancer, high grade endometrial carcinoma, and/or primary peritoneal carcinoma fallopian tube carcinoma epithelial ovarian cancer; Organization/blood samples confirmed HRD positive;
* ECOG score: 0-1;
* before, during, and after treatment of blood and tissue samples can get, and the participants agreed to at the center of the blood and tissue samples to laboratory for the expansion of the trial research purposes.
* At least one measurable lesions, CT/MRI according to RECIST 1.1 standard; • • Expectations alive at least 3 months;
* By professional gynecological oncologist judgment cannot achieve R0 reduced tumor or cannot tolerate surgery patients, cannot achieve the judgment standard of R0 reduced tumor including but not limited to:

  * Fagotti cavity mirror scoring eight points or more; 2) when the laparoscopic evaluation methods is difficult to implement, can be used on abdominal CT score 3 points or more;
  * Can't tolerate surgery judgment standard may be considered: age: the age of 70 or higher; Body mass index (BMI) : BMI 40.0 or higher; A variety of chronic diseases; Malnutrition or hypoalbuminemia; To a large number of ascites; A new diagnosis of venous thromboembolism (greater than 12 weeks of survival);
* Main organs function within 7 days before the treatment, meet the following criteria: hematologic studies: 90 g/L or higher hemoglobin, white blood cells or 3 x 109 / L, neutrophil count (ANC) absolutely acuity 1.5 x 109 / L, platelets or 90 x 109 / L; Kidney: serum creatinine < 1.5 mg/dl, glomerular filtration rate (GFR) or greater 50 ml/min (based on the screening of Fairview Laboratories formula); Liver: AST, ALT, and alkaline phosphatase (agency 3 times normal limit, total bilirubin < 1.5 times that of the upper limit of normal; Lung function: resting state oxygen saturation under 90% or more; Heart function: by echocardiography, MUGA or cardiac magnetic resonance imaging (MRI) of 40% or more LVEF; There was no electrocardiographic evidence of uncontrolled angina, severe uncontrolled ventricular arrhythmias, or acute ischemia or active conduction system abnormalities;
* Two months without obstruction history;
* Childbearing age patients effective birth control measures should be taken;
* Subjects were willing to join in this study, and sign the informed consent (ICF);
* Expected, adherence to the good curative effect and adverse reaction will be effected according to the plan calls for follow-up.

Exclusion Criteria:

* Patients who have received drugs or other cell immunotherapy in other clinical trials within 28 days before the screening period;
* Patients who have had other malignant tumors in the past 5 years;
* Acute illnesses are ongoing, or severe illnesses have occurred in the past 2 years, such as patients with active infections or fever, cardiovascular diseases (Grade III or IV heart failure), mental health issues (such as alcoholism, drug abuse);
* History of immunodeficiency, including HIV-positive status or other acquired, congenital immunodeficiency diseases;
* Organ transplant or organ failure patients, patients receiving immunosuppressive therapy after organ transplantation, or patients taking immunosuppressive drugs long-term;
* Thromboembolic events such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis, and pulmonary embolism within 6 months;
* Known allergy to any component of the final product of METR-NK preparation, including human serum albumin;
* Breastfeeding during the screening period or female subjects with positive serum or urine pregnancy tests;
* Patients with mental illnesses, including epilepsy, dementia, severe depression, bipolar disorder, etc.;
* Other conditions deemed unsuitable for inclusion by the investigator.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | 3-month
  the percentage of patients received R0 resection after METR-NK cells as neoadjuvant therapy for advanced epithelial ovarian cancer

SECONDARY OUTCOMES:
Overall Response Rate (ORR) After Neoadjuvant treatment | 3-month
Pathological complete remission rate | 3-month
Disease control rate | 3-month
Progression free survival | 2-years
Survival rate | 3-years
Adverse event | 3-month

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Cancer Hospitail, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://kchealth.com.cn/page/qywh.html